CLINICAL TRIAL: NCT05470829
Title: A Multiple-center,Randomized,Double-blind,Placebo-controlled,Multiple-dose Study Among Chinese Healthy Subjects and Chronic Hepatitis B Patients to Evaluate Safety,Tolerability,Pharmacokinetics and Preliminary Pharmacodynamics of ZM-H1505R
Brief Title: A Multiple-dose Study in Chinese Subjects to Evaluate Safety,Tolerability,PK and PD of ZM-H1505R
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Zhimeng Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZM-H1505R-102
Record Dates: First submitted 2022-07-18; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers; Hepatitis B, Chronic
Keywords: Hepatitis B, Chronic; randomized; double-blind; placebo-controlled; phase Ib
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 75mg ZM-H1505R or placebo (Experimental): 75 mg was selected for PK bridging.Twelve healthy subjects were enrolled,of which 8 subjects received ZM-H1505R and 4 subjects received placebo.
  Subjects were administrated in the morning under fasting conditions on Day 1 and afterwards Day 4 - Day 14 once daily,i.e. after 3-day washout period and followed by 11-day consecutive administration.Safety and tolerability evaluation was performed on Day 3,Day 6,Day 10 and Day 17 after the initial administration.
  Two sentinel subjects (one male and one female) were enrolled to reveived ZM-H1505R.When safety evaluation on Day 3 showed that ZM-H1505R could be tolerated by sentinel subjects,and study drug concentration of sentinel subjects after the initial administration had been analysed so that PK sampling timepoints for the remaining subjects was determined, the remaining 10 subjects were enrolled to receive ZM-H1505R or placebo at a 3:2 ratio in a randomized manner.
  Interventions: Drug: ZM-H1505R; Other: ZM-H1505R Placebo
- Cohort 1 of Part 2 50mg ZM-H1505R or placebo (Experimental): Subjects were enrolled in sequence from 50 mg dose group (cohort 1). Dose ascending was continued when safety evaluation on Day 8 showed that the lower dose could be tolerated.
  Ten chronic hepatitis B virus-infected patients were enrolled in each cohort to receive ZM-H1505R (n=8) or placebo (n=2).
  Subjects in all cohorts were administrated on Day 1 - Day 28 once daily (consecutive 28-day administration) in the morning under fasting conditions.
  Two sentinel subjects were enrolled in each cohort to reveived ZM-H1505R. When safety evaluation on Day 3 showed that ZM-H1505R could be tolerated by sentinel subjects, the remaining 8 subjects including HBeAg-positive and HBeAg-negative patients at a ratio of 4:4 were enrolled to receive ZM-H1505R or placebo at a 3:1 ratio in a randomized manner.
  Interventions: Drug: ZM-H1505R; Other: ZM-H1505R Placebo
- Cohort 2 of Part 2 100mg ZM-H1505R or placebo (Experimental): Subjects were enrolled in sequence from 100 mg dose group (cohort 2). Dose ascending was continued when safety evaluation on Day 8 showed that the lower dose could be tolerated.
  Ten chronic hepatitis B virus-infected patients were enrolled in each cohort to receive ZM-H1505R (n=8) or placebo (n=2).
  Subjects in all cohorts were administrated on Day 1 - Day 28 once daily (consecutive 28-day administration) in the morning under fasting conditions.
  Two sentinel subjects were enrolled in each cohort to reveived ZM-H1505R. When safety evaluation on Day 3 showed that ZM-H1505R could be tolerated by sentinel subjects, the remaining 8 subjects including HBeAg-positive and HBeAg-negative patients at a ratio of 4:4 were enrolled to receive ZM-H1505R or placebo at a 3:1 ratio in a randomized manner.
  Interventions: Drug: ZM-H1505R; Other: ZM-H1505R Placebo
- Cohort 3 of Part 2 200mg ZM-H1505R or placebo (Experimental): Subjects were enrolled in sequence from 200 mg dose group (cohort 3). Ten chronic hepatitis B virus-infected patients were enrolled in each cohort to receive ZM-H1505R (n=8) or placebo (n=2).
  Subjects in all cohorts were administrated on Day 1 - Day 28 once daily (consecutive 28-day administration) in the morning under fasting conditions.
  Two sentinel subjects were enrolled in each cohort to reveived ZM-H1505R. When safety evaluation on Day 3 showed that ZM-H1505R could be tolerated by sentinel subjects, the remaining 8 subjects including HBeAg-positive and HBeAg-negative patients at a ratio of 4:4 were enrolled to receive ZM-H1505R or placebo at a 3:1 ratio in a randomized manner.
  Interventions: Drug: ZM-H1505R; Other: ZM-H1505R Placebo

INTERVENTIONS:
Drug: ZM-H1505R — Part 1 dosage form:75mg dosage:Tablet frequency: Quaque die duration: Day1; Day 4~ Day 14
  Cohort 1 of Part 2 dosage form:50mg dosage:Tablet frequency: Quaque die duration: Day 1~ Day 28
  Cohort 2 of Part 2 dosage form:100mg dosage:Tablet frequency: Quaque die duration: Day 1~ Day 28
  Cohort 3 of Part 2 dosage form:200mg dosage:Tablet frequency: Quaque die duration: Day 1~ Day 28
Other: ZM-H1505R Placebo — Part 1 dosage form:75mg dosage:Tablet frequency: Quaque die duration: Day1; Day 4~ Day 14
  Cohort 1 of Part 2 dosage form:50mg dosage:Tablet frequency: Quaque die duration: Day 1~ Day 28
  Cohort 2 of Part 2 dosage form:100mg dosage:Tablet frequency: Quaque die duration: Day 1~ Day 28
  Cohort 3 of Part 2 dosage form:200mg dosage:Tablet frequency: Quaque die duration: Day 1~ Day 28

SUMMARY:
This phase Ib study included two parts in which Part I was to evaluate the safety and bridge for PK among healthy Chinese subjects and Part II were about study among Chinese chronic hepatitis B virus-infected patients. Study of Part II was carried out following the safety assessment and racial difference evaluation in Part I.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multiple-dose phase Ib study.

It aimed in this study to evaluate the safety and tolerability and to characterize the pharmacokinetics of ZM-H1505R among Chinese healthy subjects following single and multiple doses administration, and to assess whether there are ethnic differences in PK characteristic among Chinese and American healthy subjects. Study was also conducted to evaluate the safety and tolerability, to characterize the pharmacokinetics and to assess the preliminary pharmacodynamics of ZM-H1505R following multiple ascending dose administration among chronic hepatitis B virus-infected patients; the PK/PD model was established among adults to provide a basis for the oral doses determination in subsequent clinical studies of ZM-H1505R.

Part I: Study among healthy subjects for safety evaluation and PK bridging Based on the PK results among American healthy subjects in Phase Ia study, 75 mg (cohort 1) was selected for PK bridging. Twelve healthy subjects were enrolled, of which 8 subjects received ZM-H1505R and 4 subjects received placebo.

Part II: Study among chronic hepatitis B virus-infected patients Subjects in four cohorts (scheduled as cohort 2, 50 mg; cohort 3, 100 mg; cohort 4, 200 mg; cohort 5, 300 mg) were enrolled in sequence from 50 mg dose group (cohort 2). Dose ascending was continued when safety evaluation on Day 8 showed that the lower dose could be tolerated. Based on the results of PK and tolerability and PD, dose ascending to 300 mg dose group (cohort 5) from 200 mg dose group (cohort 4) was discontinued determined by sponsor and investigators. Ten chronic hepatitis B virus-infected patients were enrolled in each cohort to receive ZM-H1505R (n=8) or placebo (n=2).

ELIGIBILITY:
Inclusion Criteria:

* Able to sign Inform Consent Forms before study, and fully understand the study contents, process and potential adverse reactions;
* Able to complete the study in compliance with the protocol;
* Subjects (including their partners) agreed to adopt effective contraceptive measurements from screening to 6 months after the last administration.

Part I Proprietary:

* Male and female subjects between 18 and 50 years of age, inclusive;
* At least 50 kg for male subjects, 45 kg for female, with a Body Mass Index (BMI) between 18-28 ;
* Normal or abnormal but of no clinical significance results for physical examination and vital signs.

Part II Proprietary::

* Male and female subjects between 18 and 65 years of age, inclusive;
* At least 50 kg for male subjects, 45 kg for female subjects, with a Body Mass Index (BMI) between 18-35 kg/m2, inclusive, BMI = weight (kg) / height 2 (m2);
* Any proof of HBV infection more than 6 months (including outpatient/inpatient medical records, HBV DNA, HBsAg test sheets, etc.); or with IgM HBcAb negative and HBsAg positive at screening;
* No history of therapy including interferon/nucleoside or analog at screening, or discontinuation for more than 1 year from interferon therapy or more than 6 months from nucleoside analog therapy;
* HBV DNA ≥ 2×105 IU/mL for HBeAg-positive patients and HBV DNA ≥ 2×104 IU/mL for HBeAg-negative patients at screening;
* Serum ALT lower than 5×upper limit of normal at screening.

Exclusion Criteria:

* Major trauma or surgery within 3 months before screening;
* History of treatment that may interfere with drug absorption (e.g, subtotal gastrectomy);
* Blood donation or massive blood loss (> 450 mL) within 3 months prior to screening;
* Any history of allergy suspected to be due to any component of the study drug, or allergic constitution (allergy to multiple drug and food);
* A history of narcotic drugs intake or alcohol abuse ;
* Acute infection within 2 weeks before screening;
* Suffering from serious diseases of the circulatory, respiratory, urinary, vascular, endocrine, immune, mental and nervous systems;
* History of myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass grafting, heart failure of grade III or IV, or stroke within 6 months prior to screening;
* Patients with existing malignant tumors (except for skin non-melanoma, cervical intraepithelial neoplasia, thyroid tumor, breast tumor, etc. after treatment with no signs of recurrence);
* Any surgery or hospitalization anticipated during the study;
* Treatment history of immunosuppressants, immunomodulators (thymosin) and cytotoxic drugs within 6 months before study administration;
* Medication history of definitely strong CYP3A4 inhibitors or inducers within 2 weeks before screening;
* Involved in any other study drug administration or clinical study of medical devices within 1 month before screening; Involved in any clinical study of HBV virus nucleocapsid inhibitors in the past;
* Any abnormality of electrocardiogram not suitable for the study judged by physician;
* Positive pregnancy test results or subject is lactating for female subjects;
* Positive test results of HCV-Ab, HCV core antigen and HCV RNA (PCR); or HIV antibody; or Treponema pallidum antibody further confirmed by rapid plasma reagin (RPR) test;
* Consumption of chocolate or any diets containing caffeine or rich in xanthine, or any alcohol-containing products within 48 h before the initial administration;
* Positive results of drug abuse tests (morphine, marijuana) or alcohol breath tests;
* Other conditions in which subjects are not suitable for the study in the opinion of investigators.

Part I Proprietary:

* More than 5 cigarettes everyday within 1 month before the study;
* Intake of any prescription or over-the-counter (OTC) drugs, vitamin, herbs, other inappropriate diet or supplements in opinion of investigators within 7 days before screening;
* Positive HBsAg test results;
* Any clinically significant abnormalities in laboratory tests.

Part II Proprietary :

* Estimated glomerular filtration rate (eGFR) ˂ 60 mL/min/1.73 m2 based on serum creatinine and formula for modification of diet in renal disease (MDRD) based on values at screening;
* Patients with clinically significant acute or chronic liver disease not caused by HBV infection (including but not limited to alcoholic liver disease, severe or higher non-alcoholic fatty liver disease, autoimmune liver disease, Gilbert syndrome or other hereditary liver disease, drug-induced liver disease, etc. );
* Liver cirrhosis at clinical consideration or/and liver stiffness measurements (LSM) ≥ 12.4 kPa (for patients with ALT greater than the upper limit of normal, LSM ≥ 17.5 kPa); 27) Patients with clinically significant cardiac arrhythmias; history of risk factors for Torsade de Pointes (TdP) syndrome;
* Uncontrolled hypertension with systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg at screening;
* Patients with type I diabetes, or with newly diagnosed or poorly controlled type II diabetes (HbA1c > 8.5%);
* Left ventricular ejection fraction < 50%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ZM-H1505R among Chinese healthy subjects | 42 days
  12 healthy subjects with Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatmen
Pharmacokinetics indicators | 42 days
  PK parameters of plasma ZM-H1505R in 12 healthy subjects
Pharmacodynamics indicators | 56 days
  PK parameters of plasma ZM-H1505R in 30 chronic hepatitis B virus-infected patients
To evaluate the safety and tolerability of ZM-H1505R among chronic hepatitis B virus-infected patients | 56 Days
  30 chronic hepatitis B virus-infected patients with Abnormal Laboratory Values and/or Adverse Events That Are

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Principal Investigator — The First Hospital of Jilin University; Yanhua Ding, Principal Investigator — The First Hospital of Jilin University; Hongxin Piao, Principal Investigator — Yanbian University Affiliated Hospital (Yanbian Hospital)
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jia H, Mai J, Wu M, Chen H, Li X, Li C, Liu J, Liu C, Hu Y, Zhu X, Jiang X, Hua B, Xia T, Liu G, Deng A, Liang B, Guo R, Lu H, Wang Z, Chen H, Zhang Z, Zhang H, Niu J, Ding Y. Safety, tolerability, pharmacokinetics, and antiviral activity of the novel core protein allosteric modulator ZM-H1505R (Canocapavir) in chronic hepatitis B patients: a randomized multiple-dose escalation trial. BMC Med. 2023 Mar 16;21(1):98. doi: 10.1186/s12916-023-02814-w. PMID 36927420